CLINICAL TRIAL: NCT04254523
Title: Programmed Intermittent Bolus Versus Continuous Infusion for Epidural Analgesia in Major Abdominal Surgery: a Randomized Clinical Trial
Brief Title: Programmed Intermittent Bolus Versus Continuous Infusion for Epidural Analgesia in Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Esther Breton, Doctor Esther Breton, MD, FRCPC, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020-4832
Record Dates: First submitted 2020-01-22; First posted 2020-02-05 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Analgesia, Epidural; Pain, Postoperative
Keywords: Anesthesia, Epidural; Postoperative Period; Analgesia, Patient-Controlled
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Programmed intermittent epidural bolus (PIEB) (Experimental): Programmed intermittent epidural boluses of bupivacaine 0,1% are administered every hour.
  Interventions: Device: Programmed intermittent epidural bolus (PIEB) of bupicavaine; Device: Continuous epidural infusion (CEI) of morphine
- Continuous epidural infusion (CEI) (Experimental): A continuous epidural infusion of bupivacaine 0,1% is administered at a prescribed rate in milliliters per hour.
  Interventions: Device: Continuous epidural infusion (CEI) of bupivacaine; Device: Continuous epidural infusion (CEI) of morphine

INTERVENTIONS:
Device: Programmed intermittent epidural bolus (PIEB) of bupicavaine — Programmed intermittent epidural boluses of bupivacaine 0,1% are administered every hour. Protocolized adjustments of the dose are performed in order to obtain adequate analgesia. Standardized patient-controlled epidural boluses are available as top-ups.
  Arms: Programmed intermittent epidural bolus (PIEB)
Device: Continuous epidural infusion (CEI) of bupivacaine — A continuous epidural infusion of bupivacaine 0,1% is administered at a prescribed rate. Protocolized adjustments of the dose are performed in order to obtain adequate analgesia. Standardized patient-controlled epidural boluses are available as top-ups.
  Arms: Continuous epidural infusion (CEI)
Device: Continuous epidural infusion (CEI) of morphine — A morphine infusion (0,1mg/ml) is administered in both groups at a prescribed rate. Protocolized adjustments of the dose are performed in order to obtain adequate analgesia.

SUMMARY:
Epidural analgesia is an efficient way to relieve pain after major abdominal surgery. Two different protocols are used to provide analgesia: continuous epidural infusion (CEI) and programmed intermittent boluses (PIEB). CEI consists in the delivery of a continuous administration of the intended hourly dose. PIEB consists in the administration of sequential high pressure boluses of the intended dose. Although some studies in the postoperative setting have observed that PIEB reduces the total dose needed to ensure adequate pain control, the clinical value of this finding is still uncertain. Moreover, nursing and medical interventions to the epidural infusion rates are frequently needed in the first 48 postoperative hours to optimize the provision of analgesia. These interventions add to the already important nursing workload associated with major abdominal surgery, and are correlated with suboptimal analgesia for the patient.

This randomized controlled trial aims to compare the effect of epidural PIEB on the workload as a reflection of adequate analgesia compared to the standard CEI protocol in use. The investigators hypothesize that the use of PIEB decreases the number of interventions needed to obtain adequate analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older)
* Major abdominal surgery in an elective setting
* Thoracic epidural (between T7 and T12)

Exclusion Criteria:

* Contraindication to bupivacaine
* Contraindication to morphine
* Decision to keep the patient intubated and sedated at the end of the surgery
* Chronic opioid use (> 3 months)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-05-23 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Number of epidural infusion adjustments | 48 hours after reaching the discharge criteria from the post-anesthesia care unit (or until the beginning of the epidural weaning period, if started in less than 48 hours)
  Number of epidural infusion adjustments by the nursing team (based on the usual protocol of our institution) will be recorded.

SECONDARY OUTCOMES:
Quality of analgesia | 48 hours after reaching the discharge criteria from the post-anesthesia care unit (or until the beginning of the epidural weaning period, if started in less than 48 hours)
  Pain is measured using the numeric rating scale (NRS : 0-10, 10 being the worst possible pain).
Additional analgesia | 48 hours after reaching the discharge criteria from the post-anesthesia care unit (or until the beginning of the epidural weaning period, if started in less than 48 hours)
  Prescribed additional analgesia (IV/PO/S/C opioids or other) administered to the patient while epidural analgesia is still provided.
Incidence of hypotension | 48 hours after reaching the discharge criteria from the post-anesthesia care unit (or until the beginning of the epidural weaning period, if started in less than 48 hours)
  Documented by medical records review (vitals, medication received, temporary interruption of the local anesthetic epidural infusion, IV fluids, etc.).
Vasopressor use | 48 hours after reaching the discharge criteria from the post-anesthesia care unit (or until the beginning of the epidural weaning period, if started in less than 48 hours)
  The use of vasopressor is documented by review of the medical records.
Total epidural dose of local anesthetic administered | 48 hours after reaching the discharge criteria from the post-anesthesia care unit (or until the beginning of the epidural weaning period, if started in less than 48 hours)
  Total epidural dose of local anesthetic administered (including additional boluses ordered by the anesthesiologist and PCEA).
Total epidural dose of opioid administered | 48 hours after reaching the discharge criteria from the post-anesthesia care unit (or until the beginning of the epidural weaning period, if started in less than 48 hours)
  Total epidural dose of opioid administered.
Number of patient-controlled epidural analgesia (PCEA) administered/refused | 48 hours after reaching the discharge criteria from the post-anesthesia care unit (or until the beginning of the epidural weaning period, if started in less than 48 hours)
  Number of PCEA administered/refused.
ICU length of stay | From the admission to the ICU until the end of the ICU stay (or until the patient has met ICU discharge criteria).
  ICU length of stay
Time to postoperative mobilization | 48 hours after reaching the discharge criteria from the post-anesthesia care unit (or until the beginning of the epidural weaning period, if started in less than 48 hours)
  Time to postoperative mobilization as defined as a patient who can tolerate standing without symptoms that limit the mobilization.
Incidence of Nausea and vomiting | 48 hours after reaching the discharge criteria from the post-anesthesia care unit (or until the beginning of the epidural weaning period, if started in less than 48 hours)
  Nausea and vomiting
Incidence of Pruritus | 48 hours after reaching the discharge criteria from the post-anesthesia care unit (or until the beginning of the epidural weaning period, if started in less than 48 hours)
  Pruritus
Motor blockade | 48 hours after reaching the discharge criteria from the post-anesthesia care unit (or until the beginning of the epidural weaning period, if started in less than 48 hours)
  Bromage score is used to monitor motor blockade.
Incidence of epidural removal | 48 hours after reaching the discharge criteria from the post-anesthesia care unit (or until the beginning of the epidural weaning period, if started in less than 48 hours)
  Incidence of epidural catheter intentionally or unintentionally withdrawn.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Breton, MD, FRCPC, Principal Investigator — CHU de Québec-Universite Laval
Locations (1):
- CHU de Quebec-Universite Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: No